CLINICAL TRIAL: NCT04065698
Title: An Open-label, Single Dose, Three Sequence Study in Healthy Adult Volunteers to Evaluate the Pharmacokinetics, Safety and Tolerability of RV521 Administered as the Drug in Capsule Formulation in the Fed State and the Dry Powder Blend Formulation Dispersed in Water in the Fed and Fasted States
Brief Title: Pharmacokinetics and Safety of RV521 Formulations
Acronym: C19007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REVC005; 2019-000976-40 (EudraCT Number)
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — sisunatovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RV521 (Experimental): Three single 200 mg oral doses of RV521 administered on Day 1, Day 5 and Day 9 as either the drug in capsule (1 dosing occasion) or the dry powder blend dispersed in water (2 dosing occasions)
  Interventions: Drug: RV521

INTERVENTIONS:
Drug: RV521 — Single doses of RV521 administered as the drug in capsule formulation when fed and as the dry powder blend formulation dispersed in water when fed and whilst fasting, each on a separate dosing day.
  Other Names: Sisunatovir

SUMMARY:
The main aims of the study are to assess the pharmacokinetics and safety of single doses of RV521 administered as two different formulations

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with protocol defined contraception requirements
* In good health with no history of major medical conditions
* A body mass index (BMI) of 18-25 kg/m^2, inclusive

Exclusion Criteria:

* Evidence of any clinically significant or currently active major medical condition
* Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening
* Not willing to comply with protocol defined restrictions for intake of drugs of abuse, alcohol, nicotine-containing products, medication (prescription, OTC, herbal, vitamins/minerals etc) and specified food and drink products

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Time to maximum plasma concentration (tmax) for RV521 | Baseline to study day 11
Terminal half life (t1/2) for RV521 | Baseline to study day 11
Maximum observed plasma concentration (Cmax) for RV521 | Baseline to study day 11
Area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC0-t) for RV521 | Baseline to study day 11
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) for RV521 | Baseline to study day 11

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events as assessed by CTCAE V5.0 | Screening to final study visit (performed at 7 days following the last dose of any intervention)
Proportion of subjects with clinically significant changes in laboratory safety tests (haematology, chemistry, coagulation and urinalysis) | Screening to final study visit (performed at 7 days following the last dose of any intervention)
Proportion of subjects with morphological and/or rhythm abnormalities on ECG | Screening to final study visit (performed at 7 days following the last dose of any intervention)
Proportion of subjects with clinically significant changes in ECG time intervals (PR, QRS, QT and QTc intervals) | Screening to final study visit (performed at 7 days following the last dose of any intervention)
Proportion of subjects with clinically significant changes in vital signs (systolic blood pressure, diastolic blood pressure and pulse rate) | Screening to final study visit (performed at 7 days following the last dose of any intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lorch, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.